CLINICAL TRIAL: NCT03931733
Title: The Impact of a Receptive Music Therapy Intervention on Physiologic Measures, Pain and Agitation of Mechanically Ventilated Patients in the ICU
Brief Title: The Impact of Receptive Music Therapy in the ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 18-3129
Record Dates: First submitted 2018-12-19; First posted 2019-04-30 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Patients are assigned to either the intervention or control group based on flipping a coin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Therapy Intervention (Active Comparator): Receiving one thirty minute music therapy intervention.
  Interventions: Other: Music Therapy
- Usual Care (No Intervention): Receiving usual care for a patient in the ICU during a 30 minute intervention.

INTERVENTIONS:
Other: Music Therapy — Single thirty minute receptive music therapy intervention.
  Arms: Music Therapy Intervention

SUMMARY:
The purpose of this study is to determine whether Music Therapy has an effect on pain, agitation, and vital signs of patients in the Intensive Care Unit (ICU) when compared to usual care. Music Therapy is an intervention provided to patients after a referral by a nurse or attending physician. Patients will be assigned to two groups. The intervention group will receive 1 30 minute music therapy intervention provided by a Board Certified Music Therapist (MT-BC). The music therapy intervention will consist of a relaxation experience with live music presented by the MT-BC on an acoustic guitar, and include improvised music and/or structured songs, created as an ongoing musical experience in response to the immediate needs of the patient. Vital signs, pain, and agitation are collected pre and post. Patients assigned to the control group will receive usual care for a patient in the ICU. Vital signs, pain, and agitation will be collected.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater
* On a Mechanical Ventilator

Exclusion Criteria:

* Airborne and Special Contact Isolation
* Non English or Spanish Speaking LARs
* Pregnant
* Prisoners
* Brain Dead
* Unstable bradycardia or hypotension
* Patients who have been referred to music therapy with a goal of stimulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Change in heart rate | 30 minutes
  Physiologic Intervention
Change in respiratory rate | 30 minutes
  Physiologic Intervention
Change in Oxygenation | 30 minutes
  Physiologic Intervention

SECONDARY OUTCOMES:
Critical Care Pain Observation Tool (CPOT): Range of 0-8 Includes 2 points for: Facial expression, body movements, muscle tension, compliance with the ventilator/vocalization. Intent is decrease in pain level. | 30 minutes
  Pain
RASS: The Richmond Agitation and Sedation Scale (RASS) 0 (Alert and Calm) -1 -5: Drowsy/Unarousable +1-+4 Agitated/Combative Intent is decrease in agitation level | 30 minutes
  Agitation

CONTACTS AND LOCATIONS:
Locations (1):
- Inova Loudoun Hospital, Leesburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: No